CLINICAL TRIAL: NCT05046873
Title: A Study to Investigate the Pharmacokinetics of Semaglutide and NNC0480-0389 When Subcutaneously Administered as a Co-formulation or as Separate Injections in Healthy Participants
Brief Title: A Research Study Looking Into Blood Levels of Semaglutide and NNC0480-0389 When Given in the Same Injection or in Two Separate Injections in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9389-4679; U1111-1266-0502 (Other: World Health Organization (WHO)); 2021-001397-36 (EudraCT Number)
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0480-0389 + semaglutide(co-formulation)and placebo (Experimental): Sequence A: The participants will be administered a single subcutanous (s.c.) dose of 0.5 mg semaglutide and 5 mg NNC0480 0389 on two separate dosing visits separated by at least 8 weeks. The two drugs will be administered as a co-formulation by a single injection and a placebo injection
  Interventions: Drug: Co-formulation NNC0480 0389+Semaglutide A 10/1 mg/mL; Drug: semaglutide 1.34 mg/mL (placebo)
- NNC0480-0389 + semaglutide (separate injections) (Active Comparator): Sequence B: The participants will be administered 0.5 mg semaglutide and 5 mg NNC0480 0389 as an subcutaneus injection (s.c) on two separate dosing visits separated by at least 8 weeks. The two drugs will be administered as two separate injections.
  Interventions: Drug: Semaglutide 1.34 mg/mL; Drug: NNC0480-0389 A 10 mg/mL

INTERVENTIONS:
Drug: Co-formulation NNC0480 0389+Semaglutide A 10/1 mg/mL — Participants will receive a subcutaneus (s.c) co-formulation injection of 0.5 mg semaglutide and 5 mg NNC0480-0389 together with a subcutaneus injection (s.c) of semaglutide(placebo)on two separate dosing visits separated by at least 8 weeks.
  Arms: NNC0480-0389 + semaglutide(co-formulation)and placebo
Drug: semaglutide 1.34 mg/mL (placebo) — Participants will receive a subcutaneus (s.c) co-formulation injection of 0.5 mg semaglutide and 5 mg NNC0480-0389 together with a subcutaneus injection (s.c) of semaglutide(placebo)on two separate dosing visits separated by at least 8 weeks.
  Arms: NNC0480-0389 + semaglutide(co-formulation)and placebo
Drug: Semaglutide 1.34 mg/mL — The participants will be receive a subcutaneus (s.c) injection of 0.5 mg semaglutide and 5 mg NNC0480 0389 on two separate doing visits separated by at least 8 weeks.
  Arms: NNC0480-0389 + semaglutide (separate injections)
Drug: NNC0480-0389 A 10 mg/mL — The participants will be receive a subcutaneus (s.c) injection of 0.5 mg semaglutide and 5 mg NNC0480 0389 on two separate doing visits separated by at least 8 weeks.
  Arms: NNC0480-0389 + semaglutide (separate injections)

SUMMARY:
In this study, participants will receive semaglutide and NNC0480-0389 together at the same time. Semaglutide is a medicine that can already be prescribed, whereas NNC0480-0389 is a new potential medicine. Giving the medicines at the same time will be investigated once by using two separate syringes and once by using only one syringe containing both medicines ("co-formulation"). The co-formulation will be given together with an injection of placebo. Both medicines are tested for the treatment of type 2 diabetes. Giving the two complementary medicines at the same time is intended to lower blood sugar in people with type 2 diabetes. NNC0480-0389, in combination with semaglutide, is already being investigated in an ongoing human clinical study.

The aim of this study is to compare the amount of medicine (semaglutide and NNC0480-0389) in the blood: after participants received the medicines at the same time (0.5 mg semaglutide and 5 mg NNC0480-0389) using only one syringe (co-formulation)after participants received the medicines separately using two syringes.

For this purpose, the amount of semaglutide and NNC0480-0389 in the blood will be measured after participants received the medicines in co-formulation and after participants received the medicines using separate syringes. There will be two treatment periods: One period where participants receive the two medicines as two separate injections and another period where participants receive the two medicines in one injection (co-formulation), together with an injection of placebo. It will be randomly determined in which order participants will receive the 2 treatments (separate injections first or co-formulation first).

For both treatments the study medicines will be injected into a skin fold in the left and right stomach using a thin needle.Giving the medicines in the two treatment periods will take place at an interval of at least 8 weeks. The study can last for up to 19 weeks for each participant. This includes a screening period (up to 4 weeks), two treatment periods (5 weeks each) and a washout period (3 - 5 weeks). The washout period ensures that the given treatments and their effects have disappeared from the body. Participants will not receive any study medicines during this time. Participants will have 21 clinic visits. Some of the visits include overnight stays. Participants will have blood tests at every clinic visit.

For 4 visits (Visits 2, 11, 12 and 21; Day 1 and 36 of each period) participants must not have had any food or drink (water is allowed) for up to 8 hours before participantsr body weight is measured. Participants must be healthy and have a body mass index (BMI) between 20.0 and 29.9 kg/m2. If participants are a woman participants can only take part in this clinical study, if participants cannot get pregnant, for example, after menopause. A hormone test will be done to confirm this.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential (NCBP), aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 20.0 and 29.9 kg/m^2 (both inclusive).

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Glycosylated haemoglobin (HbA1c) more than or equal to 6.5 % (48 mmol/mol) at screening.
* Use of prescription medicinal products or non-prescription drugs, except routine vitamins, occasional use of paracetamol, ibuprofen and acetylsalicylic acid, or topical medication not reaching systemic circulation within 14 days before screening.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
AUC0-∞,sema,SD: Area under the semaglutide plasma concentration-time curve after a single dose | From baseline (visit 2/12, day 1, pre-dose) until completion of the assessment period (visit 11/21, day 36)
  h*nmol/L
AUC0-∞,NNC0480-0389,SD: Area under the NNC0480-0389 plasma concentration-time curve after a single dose | From baseline (visit 2/12, day 1, pre-dose) until completion of the assessment period (visit 11/21, day 36)
  h*nmol/L

SECONDARY OUTCOMES:
Cmax,sema,SD: Maximum plasma concentration of semaglutide after a single dose | From baseline (visit 2/12, day 1, pre-dose) until completion of the assessment period (visit 11/21, day 36)
  nmol/L
Cmax,NNC0480-0389,SD: Maximum plasma concentration of NNC0480-0389 after a single dose | From baseline (visit 2/12, day 1, pre-dose) until completion of the assessment period (visit 11/21, day 36)
  nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com